CLINICAL TRIAL: NCT01199627
Title: Tranexamic Acid Versus Placebo for the Reduction of Blood Loss in Total Hip Replacement Surgery - Randomized, Controlled and Double-masked Trial
Brief Title: Tranexamic Acid Versus Placebo for the Reduction of Blood Loss in Total Hip Replacement Surgery
Acronym: TXA-CRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Francisco Borja Barrachina Larraza, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TXA-CRT
Record Dates: First submitted 2010-09-07; First posted 2010-09-13 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Hip Replacement, Total
Keywords: total hip replacement; tranexamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Group A: 1st dose 15mg/kg of TXA (tranexamic acid) in 100ml saline 0.9% after the completion of regional anesthesia, and before the start of surgery.
  2nd dose: intravenous infusion over 10 minutes in 100ml of saline 0.9% at three hours after the first administration.
  Interventions: Drug: A
- B (Experimental): Group B: 1st dose: 10mg/kg of TXA (tranexamic acid) in 100ml 0.9% saline after the completion of regional anesthesia, and before the start of surgery.
  2nd dose: intravenous infusion over 10 minutes of 10mg/kg of TXA in 100ml saline 0.9% at three hours after the first administration.
  Interventions: Drug: B
- C (Placebo Comparator): Placebo
  Interventions: Drug: C

INTERVENTIONS:
Drug: A — Group A: 1st dose 15mg/kg of TXA (tranexamic acid) in 100ml saline 0.9% after the completion of regional anesthesia, and before the start of surgery.
  2nd dose: intravenous infusion over 10 minutes in 100ml of saline 0.9% at three hours after the first administration.
  Arms: A
Drug: B — Group B: 1st dose: 10mg/kg of TXA(tranexamic acid) in 100ml 0.9% saline after the completion of regional anesthesia, and before the start of surgery.
  2nd dose: intravenous infusion over 10 minutes of 10mg/kg of TXA in 100ml saline 0.9% at three hours after the first administration.
  Arms: B
Drug: C — Group C: 1st dose: intravenous infusion over 10 minutes in 100ml of 0.9% saline after the completion of regional anesthesia, and before the start of surgery.
  2nd dose: intravenous infusion over 10 minutes in 100ml of saline 0.9% at three hours after the first administration.
  Arms: C

SUMMARY:
The bleeding caused by hip replacement surgery (CRT) is an important source of demand for blood in the hospital. Tranexamic acid (TXA) is a drug that has proved useful in reducing bleeding associated with other surgeries and CRT results have been positive, but the variety of dosages difficult to evaluate the results To determine the efficacy and safety of TXA in reducing bleeding caused by surgery of total hip replacement.

PATIENTS: Patients ASA(American Society of Anesthesiologists) I-III that they are to perform hip replacement surgery and cementless unilateral total that have signed the informed consent.

Group A: 1st dose 15mg/kg of TXA in 100ml saline 0.9% after the completion of regional anesthesia, and before the start of surgery.

2nd dose: intravenous infusion over 10 minutes in 100ml of saline 0.9% at three hours after the first administration.

Group B: 1st dose: 10mg/kg of TXA in 100ml 0.9% saline after the completion of regional anesthesia, and before the start of surgery.

2nd dose: intravenous infusion over 10 minutes of 10mg/kg of TXA in 100ml saline 0.9% at three hours after the first administration.

Group C: 1st dose: intravenous infusion over 10 minutes in 100ml of 0.9% saline after the completion of regional anesthesia, and before the start of surgery.

2nd dose: intravenous infusion over 10 minutes in 100ml of saline 0.9% at three hours after the first administration.

STATISTICAL ANALYSIS Comparison of blood loss in groups and comparison of adverse events

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* ASA I-III
* No allergies tranexamic acid
* Informed consent signed by patient

Exclusion Criteria:

* Pregnancy or lactation.
* severe vascular ischemia (coronary or peripheral)
* previous venous thrombosis, pulmonary embolism or embolic disease (atrial fibrillation, active neoplastic disease)
* coagulopathy
* Chronic treatment with ASA(acetylsalicylic acid) or NSAIDs (nonsteroidal anti-inflammatory drugs) prior to surgery without suspension
* Hemoglobine <10
* moderate renal impairment (creatinine> 2)
* Cirrhosis
* contraindication to prophylaxis with enoxaparin
* Patients with a history of seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
blood loss (ml) | 4 hours
blood loss 8 hours (ml) | 8 hours
blood loss 24 hours (ml) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Borja Barrachina, MD, Principal Investigator — Osakidetza-Basque Country Health Service; Cesar Valero, MD, Study Chair — Osakidetza-Basque Country Health Service; Amanda Lopez, pharmacist, Study Chair — Osakidetza-Basque Country Health Service
Locations (1):
- Txagorritxu Hospital, Vitoria-Gasteiz, Alava, Spain